CLINICAL TRIAL: NCT02008370
Title: The Use of Exparel for Extended Pain Control in Minimally Invasive Cardiac Surgery
Brief Title: Exparel in Minimally Invasive Cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of available participants that meet criteria
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Giuseppe Trunfio, Director of Anesthesia for Cardiac Surgery, Maimonides Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-07-18
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Disease
Keywords: minimally invasive cardiac surgery; Exparel
MeSH Terms: conditions — Heart Diseases | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exparel infiltration (Experimental): Exparel infiltrated into wound and chest tube sites
  Interventions: Drug: Exparel infiltration

INTERVENTIONS:
Drug: Exparel infiltration — Exparel infiltrated into wound and chest tube sites
  Other Names: Bupivacaine

SUMMARY:
The investigators are presently using Exparel, a slow released local anesthestic, in patients undergoing minimally invasive cardiac surgery. The primary objective of this study is to assess the efficacy of EXPAREL when delivered into the thoracotomy and chest tube sites to provide prolonged postoperative analgesia in patients undergoing minimally invasive cardiac surgery. Efficacy will be assessed by: the effectiveness of analgesia as measured by the subject's overall postoperative pain scores and postsurgical analgesic use.

DETAILED DESCRIPTION:
Title of Study: Evaluation of the Efficacy of EXPAREL Delivered Into the Thoracotomy and Chest Tube Sites After Minimally Invasive Cardiac Surgery

Hypothesis: There is no difference in, the use of analgesics or the length of analgesia using Exparel infiltration when compared to regular bupivacaine.

Objectives: The investigators are presently using Exparel in patients undergoing minimally invasive cardiac surgery. The primary objective of this study is to assess the efficacy of EXPAREL when delivered into the thoracotomy and chest tube sites to provide prolonged postoperative analgesia in patients undergoing minimally invasive cardiac surgery. Efficacy will be assessed by: the effectiveness of analgesia as measured by the subject's overall postoperative pain scores and postsurgical analgesic use. The safety of EXPAREL will be assessed by the occurrence of all postsurgical adverse events and serious adverse event through Day 30.

Methodology: This is a prospective, open-label, non-randomized study evaluating the effectiveness of analgesia when using 266 mg EXPAREL delivered into the thoracotomy and chest tube sites by wide local infiltration. All patients in the study will undergo minimally invasive cardiac surgery. The total dose of EXPAREL for the thoracotomy and chest tube sites will be the same for up to 20 study subjects.: 266 mg of EXPAREL (13.3 mg/mL bupivacaine base). EXPAREL will be administered to each site. This total dose of Exparel is not to be exceeded in any subject. The thoracotomy and chest tube sites in this study will be performed immediately following surgery. Fentanyl will be the only opioid permitted intraoperatively. Post-operatively pain medications will be administered per standard of care by the anesthesia care team as needed to control the patient's pain. Patients will have access to a variety of rescue analgesics with appropriate routes of administration for breakthrough pain (e.g. opioids, acetaminophen, ketorolac, other nonsteroidal antiinflammatory drugs) in accordance with hospital standing orders for postsurgical pain management.

Subject reported pain will be recorded before surgery and at 2, 4, 8, 12, 24, 48, 72, 96, and 120 hours after the thoracotomy and chest tube site infiltration), and at a generally standard scheduled post-hospital discharge visit approximately 10±5 days after surgery. (Subjects discharged from the hospital will be contacted by telephone to record the scheduled pain assessments). Physician/healthcare professional assessed pain will be recorded when the patient is intubated and unable to communicate. Pain will also be assessed at the time of hospital discharge and at the last assessment (10±5 days) subjects also will be asked about their overall satisfaction with postsurgical analgesia Patients will also be asked to report any possible adverse events experienced since hospital discharge. If after Day 10±5 and through Day 30, the investigator is made aware of an adverse evevts that occurred during this period of time, this should also be recorded on the case report form if the investigator feels the event may be related to the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years inclusive and American Society of Anesthesiologists physical status 2-4.
* Undergoing minimally invasive cardiac surgery.
* Subjects must be physically and mentally able to participate in the study and complete all study assessments.
* Subjects must be able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the proposed components of thoracotomy and chest tube sites infiltration.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics
* Any subject whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful performance of a thoracotomy and chest tube sites infiltration.
* Any subject who in the opinion of the Investigator, might be harmed or be a poor candidate for participation in the study.
* Any subject, who in the opinion of the Investigator, is on chronic pain medicine, including large doses of nonsteroidal antiinflammatory drugs.
* Subjects who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during their participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Trunfio, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel Infiltration
Started | 7
Completed | 0
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Exparel Infiltration
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 59 [40 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Use of Analgesics
Description: The other primary endpoint of this study is the effectiveness of analgesia from the thoracotomy and chest tube site infiltrations as measured by the overall postsurgical analgesic use, (converted to morphine equivalents).
Time Frame: 5 days
Population: None of the patients completed to date 5: Lost to follow-up
Arm/Group | Exparel Infiltration
Number analyzed (Participants) | 0

2. Secondary Outcome: Patient Satisfaction
Description: Overall rating of subject satisfaction with postsurgical pain control
Time Frame: 10 days +/- 5 days
Population: Lost of follow-up.
Arm/Group | Exparel Infiltration
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Scores
Description: Subject reported surgical pain (using an 11-point numeric rating scale ).
Time Frame: First 5 post-op days
Population: Lost to follow up
Arm/Group | Exparel Infiltration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First 3 days
Arm/Group | Exparel Infiltration
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes